CLINICAL TRIAL: NCT05752240
Title: Transcranial Direct Current Stimulation of the Primary Motor Cortex to Treat Levodopa-induced Dyskinesias in Patients With Parkinson's Disease.
Brief Title: Transcranial Direct Current Stimulation of the Primary Motor Cortex to Treat Levodopa-induced Dyskinesias
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3944
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active stimulation (Experimental): Ten sessions of cathodic transcranial direct current stimulation over primary motor cortex
  Interventions: Device: Transcranial direct current stimulation
- Sham stimulation (Sham Comparator): Ten sessions of sham stimulation over primary motor cortex
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Ten sessions of transcranial direct current stimulation over primary motor cortex to treat levodopa-induced dyskinesia

SUMMARY:
The main objective of the study is to evaluate the efficacy of 10 sessions of transcranial direct current stimulation of the primary motor cortex to reduce levodopa-induced dyskinesia

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosis of idiopathic Parkinson's disease according to Movement Disorder Society (MDS) criteria and levodopa-induced dyskinesia;
* age between 30 and 80 years;
* ongoing therapy with levodopa;
* fulfillment of requirements for the application of transcranial magnetic stimulation (TMS), assessed by completion of the TMS screening questionnaire.

Exclusion Criteria:

* patients unable to give informed consent;
* cognitive impairment (MMSE ≤ 24);
* history of epilepsy;
* pregnant women.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2025-03-10 (Estimated)

PRIMARY OUTCOMES:
Reduction of dyskinesia | 15 days
  Change in the total score of part III of the Unified Dyskinesia Rating Scale (range 0-112, 112 is the worse outcome) in on motor state at the assessment made three days after the end of treatment compared with the assessment made at baseline in the groups of patients treated with tDCS and sham-stimulation, respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Flavia Torlizzi, Rome, Italy